CLINICAL TRIAL: NCT06950736
Title: Nicotinamide Riboside vs. Vitamin E for Enhancing Fertility in Advanced Maternal Age: A Randomized Parallel Trial
Brief Title: NR vs. Vitamin E in Enhancing Fertility
Acronym: NRVEERSAAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Qingling Yang, Associate Research Fellow, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QNCXTD2023017; QNCXTD2023017 (Other Grant/Funding Number: The First Affiliated Hospital of Zhengzhou University)
Record Dates: First submitted 2025-04-09; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Infertility Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NR (Experimental): experimental group: 600 mg/d of oral NR, NIAGEN for two months
  Interventions: Dietary Supplement: NR
- Vit E (Experimental): control group: 200 mg/d of oral Vitamin E for two months
  Interventions: Dietary Supplement: Vit E

INTERVENTIONS:
Dietary Supplement: NR — 600 mg/d of oral NR for two months
  Arms: NR
Dietary Supplement: Vit E — 200 mg/d of oral Vitamin E for two months
  Arms: Vit E

SUMMARY:
This randomized controlled trial enrolled women of advanced maternal age (≥35 years) undergoing ART, who were allocated to an intervention group (oral nicotinamide riboside, NR) or a control group (oral vitamin E, VitE) for a 2-month pre-ART intervention. The study systematically evaluated NR's regulatory effects on ovarian function and ART outcomes by measuring NAD+ levels in ovarian granulosa cells (GCs) and peripheral blood mononuclear cells (PBMCs), anti-Müllerian hormone (AMH) concentrations.

DETAILED DESCRIPTION:
Patients received daily oral supplementation of either nicotinamide riboside (NR, 600 mg/day) or vitamin E (200 mg/day) for two consecutive months, initiated on day 2 of the menstrual cycle. Participants were enrolled if they planned to undergo in vitro fertilization/intracytoplasmic sperm injection (IVF/ICSI) with a gonadotropin-releasing hormone (GnRH) antagonist protocol following the intervention period.

Biological Samples

Peripheral blood mononuclear cells (PBMC) were isolated from venous blood.

Follicular fluid containing granulosa cells and discarded oocytes were collected during routine oocyte retrieval procedures.

Hormonal and Ovarian Assessments

Baseline measurements: Blood samples were obtained on day 2-3 of the menstrual cycle prior to medication initiation to assess basal endocrine profiles (FSH, LH, E2, P, T, PRL) and anti-Müllerian hormone (AMH) levels.

Post-intervention measurements: Repeat hormonal evaluations and transvaginal ultrasound assessments (antral follicle count [AFC]) were performed on day 2-3 of the third menstrual cycle after two months of supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Infertile women aged between 35 and 42 years;
2. 0.1 ng/mL <= AMH <= 1.1 ng/ml;
3. Pregnancy aids who plan to perform in vitro fertilization and embryo transfer (antagonist program);
4. Bilateral ovaries are present;
5. Patients who voluntarily signed the informed consent and agreed to be followed up according to the requirements of the study protocol.

Exclusion Criteria:

1. Adenomyosis and uterine fibroids compression of uterine uterine line;
2. Untreated bilateral hydrosalpinx;
3. Uncured endometrial disease;
4. Any pregnancy occurred within 3 months before screening;
5. Patients with clinically significant abnormal cervical examination results within 3 months before screening;
6. Use of fertility regulators (such as clomiphene citrate, GnRH, metformin or oral contraceptives) within 1 month before randomization;
7. Use hormone drugs within 1 month before randomization;
8. Patients with acute infection of urinary and reproductive system;
9. Patients with major systemic diseases, endocrine or metabolic abnormalities that are not suitable to participate in this study, as judged by the investigator;
10. According to the judgment of the investigator, the presence of uterus (such as submucosal uterine fibroids, intermural uterine fibroids larger than 3 cm or smaller than 3 cm but affecting uterine cavity morphology, untreated endometrial polyps, uterine adhesions, uterine malformations, and ASRM stage Ⅲ-Ⅳ endometriosis). Patients with clinically significant ovarian (e.g., polycystic ovaries, ovarian cysts > 4 cm, inability to retrieve eggs from both or one ovary) or adnexa (e.g., hydrosalpinx) abnormalities;
11. Patients with unexplained abnormal uterine bleeding;
12. Patients with a history of ovarian, breast, uterus, hypothalamus, pituitary and other malignant tumors;
13. Receive donor egg or embryo preimplantation genetic screening/embryo preimplantation genetic diagnosis (PGS/PGD);
14. Known past or current thromboembolic disease;
15. Have a known serious mental illness or fail to understand the purpose and methods of the clinical trial, or fail to comply with the study procedures;
16. Patients with contraindications or allergic history to the use of GnRH-a, r-hFSH, hCGα, progesterone;
17. Those who are addicted to alcohol, tobacco, drugs or drug abuse;
18. Being exposed to teratogenic amounts of radiation, poisons and drugs and in the action period;
19. Patients with liver function injury, that is, serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were 2.5 times higher than the upper limit of normal values;
20. Persons who are HIV or syphilis positive;
21. Those with positive serum pregnancy tests;
22. Other reasons why the researcher considers it inappropriate to participate in the study. Suffers from a disease that is not suitable for the present assisted reproductive technology or for the present pregnancy;
23. Participants who had participated in other clinical trials within 3 months prior to screening.

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Follicle Counting | At the time of the first medication administration and on days 2-3 of the menstrual cycle during the second month of medication
  Transvaginal ultrasound was performed using the Voluson S8 color Doppler ultrasound system (GE, USA) to measure the diameter and number of follicles in both ovaries.
Serum AMH Levels | At the time of the first medication administration and on days 2-3 of the menstrual cycle during the second month of medication
  Blood samples for AMH were collected on days 2-3 of the menstrual cycle before ovarian stimulation.
Serum FSH Levels | At the time of the first medication administration and on days 2-3 of the menstrual cycle during the second month of medication
  Blood samples for FSH were collected on days 2-3 of the menstrual cycle before ovarian stimulation.
ART outcomes assessed by the number of clinically viable embryos and clinical pregnancy rates | From embryo transfer to the 14-day post-transfer clinical observation period
  number of top-quality day 3 embryos and transferable embryos ；the blastocyst formation rate；the number of clinically usable embryos；clinical pregnancy rates
Serum LH Levels | At the time of the first medication administration and on days 2-3 of the menstrual cycle during the second month of medication
  Blood samples for LH were collected on days 2-3 of the menstrual cycle before ovarian stimulation.
Serum P Levels | At the time of the first medication administration and on days 2-3 of the menstrual cycle during the second month of medication
  Blood samples for P were collected on days 2-3 of the menstrual cycle before ovarian stimulation.
Serum E2 Levels | At the time of the first medication administration and on days 2-3 of the menstrual cycle during the second month of medication
  Blood samples for E2 were collected on days 2-3 of the menstrual cycle before ovarian stimulation.
Serum Testosterone levels | At the time of the first medication administration and on days 2-3 of the menstrual cycle during the second month of medication
  Blood samples for testosterone were collected on days 2-3 of the menstrual cycle before ovarian stimulation.
Antral Follicle Count Retrived | Immedietly after oocyte retrived
  Transvaginal ultrasound was performed using the Voluson S8 color Doppler ultrasound system (GE, USA) to measure the diameter and number of follicles in both ovaries.
Oocytes Retrived | Immedietly after oocyte retrived
  Number of oocytes retrieved in Antagonist Protocol
NAD+ Levels in PBMCs | At the time of the first medication administration and on days 2-3 of the menstrual cycle during the second month of medication
  NAD+ levels and NAD+/NADH in PBMCs before and after medication
NAD+ Levels in GCs | Immedietly after oocyte retrived
  NAD+ levels and NAD+/NADH in GCs
Number of Day 3 embryos | Day 3 of Embryo Culture
  Number of Day 3 embryos
Number of Day 3 top-quality embryos | Day 3 of Embryo Culture
  embryos cultured to the third day post-fertilization that meet specific morphological criteria for optimal quality
Number of transferable embryos | Day 3 of Embryo Culture
  total number of embryos that meet predefined laboratory criteria for potential implantation
Blastocyst Formation Rate | Day 6 of Embryo Culture
  Blastocyst Formation Rate (BFR) = (Number of embryos reaching blastocyst stage ÷ Total embryos cultured to Day 5-6) × 100%

IPD SHARING:
Plan to Share IPD: No